CLINICAL TRIAL: NCT06046196
Title: A Randomized, Multicenter, Open-label, Parallel, Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of Sarpogrelate SR in Patients Having Intermittent Claudication Among Chronic Artery Occlusive Disease
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Sarpogrelate SR in Patients With Chronic Artery Occlusive Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC044
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Arterial Occlusive Diseases; Intermittent Claudication
Keywords: Sarpogrelate Sustained Release; Sarpogrelate
MeSH Terms: conditions — Arterial Occlusive Diseases; Intermittent Claudication | interventions — sarpogrelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarpogrelate SR 300mg, QD (Experimental): Sarpogrelate SR 300mg, QD
  Interventions: Drug: Sarpogrelate SR
- Sarpogrelate 100mg, TID (Active Comparator): Sarpogrelate 100mg, TID
  Interventions: Drug: Sarpogrelate

INTERVENTIONS:
Drug: Sarpogrelate SR — Sarpogrelate SR 300mg, once a daily, for 24weeks
  Other Names: Anplag SR Tab. 300mg
  Arms: Sarpogrelate SR 300mg, QD
Drug: Sarpogrelate — Sarpogrelate 100mg, 3 times a day, for 24weeks
  Other Names: Anplag Tab. 100mg
  Arms: Sarpogrelate 100mg, TID

SUMMARY:
This clinical trial aims to assess the non-inferiority of Sarpogrelate SR 300mg once daily compared to Sarpogrelate 100mg three times daily in patients having intermittent claudication among chronic artery occlusive disease, based on changes in the Ankle-Brachial Index (ABI).

DETAILED DESCRIPTION:
The clinical trial is a randomized, multicenter, open-label, parallel-group, Phase 4 study conducted to evaluate the non-inferiority of Sarpogrelate SR 300mg once daily compared to Sarpogrelate 100mg three times daily in patients having intermittent claudication among chronic artery occlusive disease. Eligible patients who sign the informed consent form voluntarily will receive the investigational products. Subsequently, they will undergo observation and various assessments at the 12-week and 24-week visits. The trial is designed to determine whether Sarpogrelate SR 300mg once daily is inferior to Sarpogrelate 100mg three times daily in terms of changes in the Ankle-Brachial Index (ABI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 19
* Diagnosis of chronic arterial occlusive disease
* Experience of intermittent claudication symptoms for at least 3 months
* Receiving Sarpogrelate for a minimum of 4 weeks prior to the baseline
* Lower limb pain measured at VAS 40mm or higher at baseline

Exclusion Criteria:

* Patients with coronary artery disease or cerebrovascular disease related to arteriosclerosis undergoing or scheduled for surgery or medication treatment
* Patients with a history of severe heart failure within the 6 months prior to the screening
* Patients with a history of bleeding
* Patients receiving anticoagulants or medications with antiplatelet activity at baseline
* Patients diagnosed with peripheral neuropathy and currently taking neuropathic pain medications
* Patients with infectious or progressive fibrotic diseases such as rheumatoid arthritis, systemic lupus erythematosus, idiopathic pulmonary fibrosis, etc

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Ankle-Brachial Index (ABI) | from baseline to the 12-week and 24-week
  To evaluate the efficacy following administration of Sarpogrelate SR

SECONDARY OUTCOMES:
Change in Lower Limb Pain Visual Analogue Scale (VAS) | from baseline to the 12-week and 24-week timepoints
  To evaluate the efficacy following administration of Sarpogrelate SR
Change in Medication Adherence Index (MMAS-8) | from baseline to the 12-week and 24-week timepoints.
  To evaluate the efficacy following administration of Sarpogrelate SR
Change in Walking Impairment Questionnaire (WIQ) | from baseline to the 12-week and 24-week timepoints
  To evaluate the efficacy following administration of Sarpogrelate SR
the Rate of subjects with grades of Spontaneous Pain, Numbness, and Coldness | at baseline, 12-week, and 24-week timepoints
  To evaluate the efficacy following administration of Sarpogrelate SR

CONTACTS AND LOCATIONS:
Overall Officials: Jungyo Gwon, Principal Investigator — Asan Medical Center
Locations (7):
- South Korea (7):
  - GangNeung Asan Hospital, Gangneung-si, Gangwon-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Korea University ANAM Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No